CLINICAL TRIAL: NCT01036568
Title: Neuroimaging Studies of Neurophysiological Phenotypes in Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906405; 06-DA-N405
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-03-07

CONDITIONS: Schizophrenia; Psychosis
Keywords: Psychosis; Smooth Pursuit; Motion Perception; Neurophysiology; fMRI
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

SUMMARY:
Background:

- Eye tracking, the ability to focus on and follow a moving target with the eyes, is often difficult for people who have schizophrenia. Research has shown that first-degree relatives of people with schizophrenia, such as parents and siblings, also tend to have difficulty with smooth eye movement and eye tracking. Researchers are interested in using functional magnetic resonance imaging (fMRI) to study brain activity during eye tracking tests in order to better understand the effect that schizophrenia has on brain function.

Objectives:

- To study eye-tracking and eye-tracking impairments in people with and without schizophrenia.

Eligibility:

- Individuals between 18 and 62 years of age in one of three groups: (1) patients who have been diagnosed with schizophrenia/schizoaffective disorder, (2) first-degree relatives of patients in group 1, and (3) healthy volunteers with no family history of psychosis.

Design:

* The study will involve two visits, one screening session and one testing session. Each session will take about 3 hours.
* Participants will be asked to avoid consuming alcohol and restrict consumption of caffeine before the start of the study. Participants will provide urine and breath samples to be tested for chemicals that may interfere with the study.
* Participants will visit the clinical center the morning of the day before the scanning session to provide blood and urine samples as required. Participants will return and be admitted for an overnight stay later that afternoon or evening.
* During the screening session, participants will provide a medical and psychological history, provide blood samples, and learn the eye movement tasks they will do during the scanning session.
* During the scanning session, participants will have an fMRI scan. During the scan, they will perform eye movement tasks that involve following moving light targets on a screen, and will also perform other tasks that test the ability to think and pay attention.

DETAILED DESCRIPTION:
Objective:

The proposed protocol aims to combine functional magnetic resonance imaging (fMRI) and SPEM eyetracking measures to study 1) the neural circuit controlling the psychophysical, cognitive, and oculomotor aspects of eyetracking; 2) the underlying neural mechanism of schizophrenia-related eyetracking impairments; and 3) the degree to which pursuit-related imaging changes aggregate in families. The human eye movement system is complex. It is likely that only components of the system, rather than the whole system, are involved in the pathology of schizophrenia.

Study Population:

Three groups of subjects will be tested: schizophrenic patients (approximately n=60), full siblings of patients (approximately n=60), and healthy controls without family history of psychosis (approximately n=60). To reach this goal of 60 per group we expect to enroll 225 subjects.

Design:

Experiments in this protocol employ fMRI in combination with psychophysical and oculomotor paradigms to dissect the neural correlates of the neurophysiological components controlling pursuit eye movement. A high-resolution in-magnet eyetracking system will be used during imaging. Using this imaging technology we will be able to associate behavioral performance with specific brain regions.

Outcome Measures:

Combining fMRI and visual neuroscience techniques, this protocol will study the functional neuroanatomic underpinnings of smooth pursuit eye movement (SPEM) deficits in schizophrenia. We aim to establish a pathophysiological model of the illness based on the SPEM paradigm. Such a disease model may provide safe in vivo examination of the effects of pharmacological interventions, comorbidity, and functionality relating to schizophrenia. For example, patients with schizophrenia have high comorbidity of nicotine use. High incidence of substance abuse in schizophrenia suggests that the two conditions may share some common pathophysiology. Excessive nicotine use in schizophrenia is increasingly viewed as a form of self-medication by patients to correct underlying pathophysiological changes caused by the illness. We have found that nicotine can transiently improve smooth pursuit eye movement deficits in patients. We are currently examining the nicotinic effect on the learning components of smooth pursuit eye movement in schizophrenic patients using fMRI. This is an example on how carefully validated behavioral/imaging paradigm can be used as a pathophysiological model in aiding the study of complex brain illness including schizophrenia and substance abuse. Clearly, this research direction also requires a parallel research effort that aims at in-depth understanding of the foundational neural mechanism of the smooth pursuit eye movement itself.

ELIGIBILITY:
* INCLUSION CRITERIA:

All Subjects:

1. must be 18-62 years of age.
2. must be in good general health based on medical history and physical examination.

Schizophrenic patients:

1. must have a DSM-IV diagnosis of schizophrenia.
2. must be clinically stable in the opinion of the patient s treating clinician with no change in antipsychotic medications or any dosage adjustment for 2 weeks or more preceding study enrollment as well as 2 weeks or more prior to the MRI scan.

Relatives of patients:

1. must be first degree relatives (full sibling, parent, or offspring)

EXCLUSION CRITERIA:

All subjects:

1. Individuals who have alcohol and/or marijuana dependence
2. Individuals who are pregnant; Urine pregnancy tests will be performed on all female volunteers of childbearing potential before each experimental session.
3. Individuals who are unable to undergo MRI scanning due to pregnancy, implanted metallic devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts) or claustrophobia.
4. Individuals who have major medical illnesses that may affect normal brain functioning or safety lying in the scanner. Examples of these conditions include, but not limited to, stroke, seizure, HIV/AIDS, uncontrolled high blood pressure, history of significant head trauma, CNS infection or tumor based on medical history, peripheral vascular diseases, coagulopathies, history of superficial or deep vein thrombosis.
5. Individuals who partake in significant alcohol or other drug use, other than nicotine dependence. Significant drug use is defined as a history of alcohol or other substance dependence in the past 6 months or current substance abuse, with the following few exceptions. Subjects may be users of alcohol and/or marijuana but may not meet criteria for dependence.
6. Individuals with significant ophthalmological and/or neurological conditions who have severe vision impairments such that they cannot follow a moving dot 60 cm in front of them are excluded. Participants with reduced vision are included as long as they can follow a moving dot 60 cm in front of them.

Healthy controls:

1. Individuals with psychiatric illness. The SCID and Structured Interview for DSM-IV Personality Diagnoses (SIDP) will be used to exclude volunteers with Axis I and II disorders.
2. Individuals with a family history of psychotic illness according to Family History Research Diagnostic Criteria (FH-RDC).

First Degree Relatives of patients:

1. First degree relatives with a DSM-IV Axis I diagnosis of psychosis, with the exception that a relative with a past history of psychosis will be included if symptoms are not present, and he/she is not taking antipsychotic drugs.
2. First degree relatives that meet SIDP criteria for an Axis II disorder with exceptions made for relatives meeting criteria for schizophrenia spectrum personality disorders (SSPD).

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2006-02-14; Study Completion 2013-03-07

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland

REFERENCES:
- [Background] Andreasen NC, Endicott J, Spitzer RL, Winokur G. The family history method using diagnostic criteria. Reliability and validity. Arch Gen Psychiatry. 1977 Oct;34(10):1229-35. doi: 10.1001/archpsyc.1977.01770220111013. PMID 911222
- [Background] Assad JA, Maunsell JH. Neuronal correlates of inferred motion in primate posterior parietal cortex. Nature. 1995 Feb 9;373(6514):518-21. doi: 10.1038/373518a0. PMID 7845463
- [Background] Avila MT, Adami HM, McMahon RP, Thaker GK. Using neurophysiological markers of genetic risk to define the boundaries of the schizophrenia spectrum phenotype. Schizophr Bull. 2003;29(2):299-309. doi: 10.1093/oxfordjournals.schbul.a007006. PMID 14552505